CLINICAL TRIAL: NCT01355952
Title: An Open-Label Pilot Trial of Alpha Lipoic Acid (ALA) for Weight Loss in Schizophrenia
Acronym: ALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Cenk Tek, Associate Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1103008158
Record Dates: First submitted 2011-05-16; First posted 2011-05-19 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Obesity; Weight Loss; Schizophrenia
Keywords: Obesity; Weight Loss; Schizophrenia; Alpha Lipoic Acid
MeSH Terms: conditions — Obesity; Weight Loss; Schizophrenia | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alpha Lipoic Acid (Experimental): taking 1800mg daily (600mg 3 times per day) Alpha Lipoic Acid (ALA) open-label for 10 weeks.
  Interventions: Dietary Supplement: Alpha Lipoic Acid

INTERVENTIONS:
Dietary Supplement: Alpha Lipoic Acid — 600mg three times per day (1800mg total) daily for 10 weeks

SUMMARY:
The aim of this study is to collect pilot data to compare the effectiveness of treatment with Alpha Lipoic Acid (ALA) for reduction in body weight in 40 obese outpatients with schizophrenia or schizoaffective disorder in an open-label pilot trial. The investigators also plan to test the feasibility of utilizing ALA as a weight loss agent for obese outpatients with schizophrenia or schizoaffective disorder in terms of tolerability, schizophrenia symptoms, cognition and side effects. We have run a total of 12 non-diabetic participants and are now recruiting diabetic patients in hopes of comparing the two groups.

DETAILED DESCRIPTION:
Design: This is a ten week open-label, fixed dose clinical study of alpha lipoic acid (ALA) for the treatment of antipsychotic weight gain in outpatients with schizophrenia or schizoaffective disorder.

Study Endpoints: The primary outcome measure is change in body weight from baseline. Secondary outcome measures are fasting serum glucose, glycosylated hemoglobin, insulin, LDL cholesterol, triglyceride levels, quality of life (Q-LES-Q), Clinical Global Impression (CGI) scores and performance on the The Brief Assessment of Cognition in Schizophrenia neurocognitive battery (BACS). (after preliminary analysis, we have changed the cognitive assessment to the DSST task only. The investigators are also going to conduct exploratory analyses of food craving, food preference and food frequency.

Subjects: Subjects will be recruited from the Psychosis Program and clinician referrals from other teams at the CMHC. Based on our previous weight loss studies the investigators expect very high enthusiasm from the subjects.

Procedure and assessment schedule: Subjects who meet the inclusion/exclusion criteria will participate in a multi-step screening process where demographic information will be gathered, weight and BMI will be measured and fasting blood will be taken, and if you are a female, a urine sample will be tested for pregnancy. If lab results are adequate, the subject will continue on to a baseline visit where they will start taking alpha lipoic acid (ALA) at 600mg three times a day (1800mg total) for a total of ten weeks. At each visit, weight will be obtained, scheduled blood will be drawn and study ratings will be conducted. A short visit with the physician every two weeks ensures safety and improves rating fidelity. Medication compliance will be ensured with pill counts, feedback and encouragement that is standard for clinical trials with schizophrenia patients. Research scales are standard schizophrenia and food scales.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years;
2. Meet DSM-IV criteria for schizophrenia or schizoaffective disorder (confirmed from clinical chart)
3. Overweight, as defined with a BMI of equal to or greater than 27 kg/m²;
4. Be on a stable dose of antipsychotic medication; i.e. at least one month with no dosage change, and two months from an antipsychotic switch;
5. Deemed to be symptomatically stable by the clinical staff in the last two months;

8) English speaking

Exclusion Criteria:

1. A history of dementia, mental retardation or other neurological disorder that may interfere with study ratings;
2. Not capable of giving informed consent for participation in this study;
3. Ongoing pregnancy;
4. A medical disorder that is known to cause obesity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | week 10
  change in body weight from baseline

SECONDARY OUTCOMES:
Change in lab values | week 10
  change in fasting serum glucose, glycosylated hemoglobin, insulin, LDL cholesterol, triglyceride levels from baseline to week 10
Change in ratings of quality of life and cognition | week 10
  change in quality of life (Q-LES-Q), Clinical Global Impression (CGI) scores and performance on the The Brief Assessment of Cognition in Schizophrenia neurocognitive battery (BACS).

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Tek, M.D., Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Ratliff JC, Palmese LB, Reutenauer EL, Tek C. An open-label pilot trial of alpha-lipoic acid for weight loss in patients with schizophrenia without diabetes. Clin Schizophr Relat Psychoses. 2015 Jan;8(4):196-200. PMID 23471087